CLINICAL TRIAL: NCT05027516
Title: An Open Label Randomized Controlled Trial Comparing the Effect of Ceftriaxone Plus Azithromycin Versus Ceftriaxone for the Treatment of Neisseria Gonorrhoeae on the Resistome
Brief Title: Trial Comparing Ceftriaxone Plus Azithromycin Versus Ceftriaxone for the Treatment of Gonorrhea
Acronym: ResistAZM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ITM202101
Record Dates: First submitted 2021-07-20; First posted 2021-08-30 (Actual); Results first posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-02

CONDITIONS: Neisseria Gonorrhoeae
MeSH Terms: interventions — Ceftriaxone; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rocephine® (Active Comparator): ceftriaxone 1g + lidocaine 35mg; intramuscular injection
  Interventions: Drug: Rocephin
- Rocephine® + Azithromycin (Active Comparator): ceftriaxone 1g + lidocaine 35mg intramuscular injection + azithromycin 2g orally
  Interventions: Drug: Rocephin; Drug: Azithromycin

INTERVENTIONS:
Drug: Rocephin — Single dose of Rocephine® (= ceftriaxone 1g + lidocaine 35mg) intramuscular injection
  Other Names: Ceftriaxone
Drug: Azithromycin — Single dose of Rocephine® (= ceftriaxone 1g + lidocaine 35mg) intramuscular injection + single dose of azithromycin 2g orally
  Other Names: Zithromax
  Arms: Rocephine® + Azithromycin

SUMMARY:
In this Randomized Controlled Trial, the investigators will recruit 42 men attending the STI and HIV clinic at the Institute of Tropical Medicine, with a diagnosis of N. gonorrhoeae and randomize them 1:1 to receive either ceftriaxone or ceftriaxone/azithromycin. They will be followed-up for a test of cure visit at day 14 post-treatment where urine, oropharyngeal and anorectal samples will be taken to test for cure and monitor treatment effects on the microbiome and resistome. The primary outcome will be evaluating the difference in the abundance of resistance conferring genes in the rectal microbiome in the two arms, 14 days after the receipt of therapy.

ELIGIBILITY:
Inclusion criteria:

1. Able and willing to provide written informed consent
2. Male sex at birth
3. At least 18 years old
4. Confirmed diagnosis of urethritis, proctitis or pharyngitis N. gonnorrhea - symptomatic or asymptomatic (Diagnosis of N. gonnorrhea will be by a positive NAAT performed according to the ITMs current laboratory protocols or for patients with urethritis a positive gram/methylene blue stain)

Exclusion criteria:

1. Use of any macrolide antibiotics (azithromycin, clarithromycin, erythromycin, roxithromycin, spiramycin) in previous 6 months
2. Known contra-indications or allergy to ceftriaxone, azithromycin or lidocaine
3. Presence of any other condition, including other Sexually Transmitted Infections that will (likely) require the administration of another antibiotic at the time of enrollment, as assessed by the treating physician

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Inclusion of male sex at birth
Enrollment: 42 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Tropical Medicine, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rocephine® | Rocephine® + Azithromycin
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rocephine® | Rocephine® + Azithromycin | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [28.5 to 41.75] | 41.5 [29.75 to 45] | 40 [29.25 to 44]
Sex/Gender, Customized [Number; unit: participants]
  Male sex at birth | 22 | 20 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
HIV status: Positive [Count of Participants; unit: Participants] | 5 | 4 | 9
HIV status: Negative [Count of Participants; unit: Participants] | 17 | 16 | 33
Symptomatic NG [Count of Participants; unit: Participants] | 7 | 6 | 13
Number of partners (last 3 months) [Median (Inter-Quartile Range); unit: partners] | 5 [3 to 6] | 5 [3.75 to 10] | 5 [3 to 8.25]
Use of antibiotics in the last 12 months [Count of Participants; unit: Participants] | 8 | 10 | 18
Amoxicillin/Clavulanic acid [Count of Participants; unit: Participants] | 0 | 2 | 2
Ceftriaxone [Count of Participants; unit: Participants] | 0 | 0 | 0
Doxycycline [Count of Participants; unit: Participants] | 0 | 0 | 0
Penicillin [Count of Participants; unit: Participants] | 0 | 0 | 0
PrEP use [Count of Participants; unit: Participants] | 14 | 13 | 27
Infection site: Anorectal [Count of Participants; unit: Participants] | 2 | 1 | 3
Infection site: Urethral [Count of Participants; unit: Participants] | 4 | 5 | 9
Infection site: Pooled [Count of Participants; unit: Participants] | 16 | 14 | 30
Teeth discoloration [Count of Participants; unit: Participants] | 0 | 0 | 0
Dental caries [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Macrolide Resistance Determinants
Description: During the bioinformatic analyses, each identified antibiotic-resistance determinant will be categorized at the class level using a read-based classification tool. The primary outcome will be the ratio of mean macrolide resistance determinants in the day 14 anorectal samples between the two treatment groups. This ratio will be calculated by dividing the mean normalized read count of macrolide- resistance determinants categorized at the class level in the Ceftriaxone/Azithromycin group by the corresponding mean quantity in the Ceftriaxone group.
Time Frame: Day 14
Population: The primary analysis of assessing the ratio between the mean normalized read count of macrolide resistance determinants in anorectal microbiome between the two groups was done using permutation test with 10 000 permutations.
Measure: Mean (95% Confidence Interval); unit: normalized determinants/million reads
Groups:
- Rocephine: Ceftriaxone 1g + lidocaine 35mg intramuscular injection on day 0
- Azithromycin / Rocephine®: ceftriaxone 1g + lidocaine 35mg intramuscular injection on day 0
  azithromycin 2g per os on day 0
Arm/Group | Rocephine | Azithromycin / Rocephine®
Number analyzed (Participants) | 22 | 20
normalized determinants/million reads | 110.3 [64.54 to 156.06] | 167.53 [97.86 to 237.19]
Statistical Analysis 1: Comparison: Rocephine vs Azithromycin / Rocephine®; Test type: Superiority; p = 0.1026, Permutation testing; Ratio = 1.05, 95% CI 2-sided [0.55 to 1.83]

2. Secondary Outcome: Read Count of Resistance Determinants for Each Non-macrolide Antibiotic Class
Description: The ratio of mean normalized read count of resistance determinants for each non-macrolide antibiotic class in the day 14 anorectal samples between the two treatment groups
Time Frame: Day 14
Population: The normalized macrolide resistance determinants were calculated by dividing the number of macrolide resistance reads by the total number of bacterial reads. The resulting proportion was then multiplied by 106 to present results in normalized determinants per million reads. No sample had a total number of reads below 95 thousand.
Measure: Mean (95% Confidence Interval); unit: normalized determinants/million reads
Groups:
- Rocephine®: ceftriaxone 1g + lidocaine 35mg intramuscular injection
- Rocephine® + Azithromycin / Rocephine®: ceftriaxone 1g + lidocaine 35mg intramuscular injection on day 0
  azithromycin 2g per os on day 0
Arm/Group | Rocephine® | Rocephine® + Azithromycin / Rocephine®
Number analyzed (Participants) | 22 | 20
normalized determinants/million reads
  Aminoglycosides | 34.41 [11.36 to 57.45] | 22.22 [14.98 to 29.46]
  Betalactams | 110.46 [80.17 to 140.76] | 89.82 [68.36 to 111.28]
  Bacitracin | 4.63 [0 to 11.21] | 1.11 [0 to 2.96]
  Glycopeptides | 0.26 [0 to 0.77] | 0.14 [0 to 0.4]
  Trimethoprim | 2.73 [0.7 to 4.77] | 1.55 [0.4 to 2.69]
  Cationic antimicrobial peptides | 16.52 [0 to 38.45] | 5.52 [0 to 14.65]
  Mupirocin | 0.84 [0 to 1.86] | 0 [0 to 0]
  Metronidazole | 0.2 [0 to 0.61] | 0.06 [0 to 0.19]
  Fluoroquinolones | 9.44 [0 to 21.97] | 23.9 [0 to 68.13]
  Sulfonamides | 5.47 [0 to 11.84] | 0.62 [0 to 1.76]
  Tetracyclines | 348.12 [286.41 to 409.82] | 423.8 [361.52 to 486.09]
Statistical Analysis 1: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For aminoglycosides; Test type: Superiority; p = 1, Permutation testing; Ratio = 1.12, 95% CI 2-sided [0.47 to 2.19]
Statistical Analysis 2: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For betalactams; Test type: Superiority; p = 1, Permutation testing; Ratio = 1.01, 95% CI 2-sided [0.69 to 1.44]
Statistical Analysis 3: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For bacitracin; Test type: Superiority; p = 1, Permutation testing; Ratio = 3.79, 95% CI 2-sided [0.05 to 20.15]
Statistical Analysis 4: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For glycopeptides; Test type: Superiority; p = 1, Permutation testing; Ratio = 0.83, 95% CI 2-sided [0 to 1.91]
Statistical Analysis 5: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For trimethoprim; Test type: Superiority; p = 1, Permutation testing; Ratio = 1.19, 95% CI 2-sided [0.32 to 3.15]
Statistical Analysis 6: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For cationic antimicrobial peptides; Test type: Superiority; p = 1, Permutation testing; Ratio = 2.82, 95% CI 2-sided [0.07 to 14.64]
Statistical Analysis 7: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For mupirocin; Test type: Superiority; p = 1, Permutation testing; Ratio = 1.49, 95% CI 2-sided [0 to 5.34]
Statistical Analysis 8: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For metronidazole; Test type: Superiority; p = 1, Permutation testing; Ratio = 1.2, 95% CI 2-sided [0 to 3.22]
Statistical Analysis 9: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For fluoroquinolones; Test type: Superiority; p = 1, Permutation testing; Ratio = 6.44, 95% CI 2-sided [0.02 to 46.02]
Statistical Analysis 10: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For sulfonamides; Test type: Superiority; p = 1, Permutation testing; Ratio = 10.6, 95% CI 2-sided [0.01 to 148.86]
Statistical Analysis 11: Comparison: Rocephine® vs Rocephine® + Azithromycin / Rocephine®; For tetracyclines; Test type: Superiority; p = 0.5621, Permutation testing; Ratio = 1.01, 95% CI 2-sided [0.79 to 1.27]

3. Secondary Outcome: Acquisition of Phenotypic Resistance to Azythromycin by N. Gonnorrhea
Description: The difference in time until acquisition of phenotypic resistance to Azithromycin by N. gonnorrhea in the morbidostat upon exposure to commensal Neisseria DNA extracts from each treatment group
Time Frame: Day 0 and Day 14
Population: change of proportion of isolates resistant to azithromycin between day 0 and day 14
Measure: Number; unit: Proportion of isolates resistant to AZM
Arm/Group | Rocephine® | Rocephine® + Azithromycin
Number analyzed (Participants) | 22 | 20
Proportion of isolates resistant to AZM
  Streptococci day 0 | 0.649 | 0.669
  Streptococci day 14 | 0.572 | 0.739
  Commensal Neisseria day 0 | 0.534 | 0.471
  Commensal Neisseria day 14 | 0.542 | 0.638
Statistical Analysis 1: Comparison: Rocephine®; For streptococci; Test type: Superiority; p = 0.196, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Rocephine® + Azithromycin; For streptococci; Test type: Superiority; p = 0.568, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Rocephine®; For Neisseria; Test type: Superiority; p = 0.978, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Rocephine® + Azithromycin; For Neisseria; Test type: Superiority; p = 0.184, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected over the whole study duration (4 months).
Arm/Group | Rocephine® | Rocephine® + Azithromycin
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 2/22 | 4/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rocephine® (N=22) | Rocephine® + Azithromycin (N=20)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
pain at injection site (General disorders) | 2 (2) | 1 (1)
presyncope (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT05027516/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT05027516/SAP_001.pdf
  • Informed Consent Form (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/16/NCT05027516/ICF_002.pdf